CLINICAL TRIAL: NCT00918658
Title: Collection of Bone Marrow and Peripheral Blood for Testing of Notch-induced Natural Killer Cell Activity
Brief Title: Study of Natural Killer Cells in Bone Marrow and Blood Samples From Patients With and Without Hematologic Cancer
Status: Terminated | Type: Observational
Why Stopped: PI closed lab
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE2Z08; P30CA043703 (NIH); CASE2Z08 (Other: Case Comprehensive Cancer Center); CASE-2Z08-CC502 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Leukemia; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: childhood chronic myelogenous leukemia; chronic myelogenous leukemia; adult acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia; adult acute myeloid leukemia; childhood acute myeloid leukemia/other myeloid malignancies; multiple myeloma
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Immunologic Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To collect normal and malignant cells in bone marrow and peripheral blood samples from patients with acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, or multiple myeloma and from patients with no malignancy to use as target cells in cytotoxicity assays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with hematologic cancer: Patients with acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, or multiple myeloma
  Interventions: Other: biologic sample preservation procedure; Other: immunologic technique; Other: laboratory biomarker analysis
- Patients without cancer: Patients who do not have cancer.
  Interventions: Other: biologic sample preservation procedure; Other: immunologic technique; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: biologic sample preservation procedure — All specimens will be collected using the Pathology Residual Tissue Procurement.
Other: immunologic technique — Information about HLA type and immunophenotype of the malignant cells is collected from the patient's medical record.
Other: laboratory biomarker analysis — Bone marrow aspirates and/or peripheral blood samples are collected and used as target cells in standard cytotoxicity assays, with notch-induced natural killer (N-NK) cells as the effector cells, to determine whether N-NK cells are capable of killing malignant cells and/or non-malignant cells. Receptor-blocking antibodies may be added to determine which NK cell receptors are responsible for malignant cell recognition and killing.

SUMMARY:
RATIONALE: Collecting and storing samples of bone marrow and blood from patients with cancer to study in the laboratory may help doctors find better ways to treat the cancer.

PURPOSE: This research study is looking at natural killer cells in bone marrow and blood samples from patients with hematologic cancer and from patients who do not have cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To collect normal and malignant cells in bone marrow and peripheral blood samples from patients with acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, or multiple myeloma and from patients with no malignancy to use as target cells in cytotoxicity assays.
* To collect information about HLA type and immunophenotype of malignant cells as determined by clinical flow cytometry.

OUTLINE: Bone marrow aspirates and/or peripheral blood samples are collected and used as target cells in standard cytotoxicity assays, with notch-induced natural killer (N-NK) cells as the effector cells, to determine whether N-NK cells are capable of killing malignant cells and/or non-malignant cells. Receptor-blocking antibodies may be added to determine which NK cell receptors are responsible for malignant cell recognition and killing.

Information about HLA type and immunophenotype of the malignant cells is collected from the patient's medical record.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * No evidence of malignancy
  * Diagnosis of one of the following:

    * Acute myeloid leukemia
    * Acute lymphoblastic leukemia
    * Chronic myelogenous leukemia
    * Multiple myeloma

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Collection of normal and malignant cells to use as target cells in cytotoxicity assays | We anticipate collecting approximately 30 samples in total, over a 1-2 year period.

CONTACTS AND LOCATIONS:
Overall Officials: Rose Beck, MD, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States